CLINICAL TRIAL: NCT05914337
Title: Investigation Into the Effects of Exercise on microRNA Expressions in Patients With Rheumatoid Arthritis
Brief Title: Exercise on microRNA in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA_miRNA
Record Dates: First submitted 2023-04-17; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; exercise; microRNA
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rheumatoid Arthritis Group (Experimental): 30 patients aged 18-60 years who met the 2010 American College of Rheumatology / European League Against Rheumatism Rheumatoid arthritis criteria were included in the study. A program consisting of strengthening and stretching exercises 2 days a week was applied to the study group for 8 weeks. One day a week, 30 minutes of mild moderate walking was requested. 30 healthy controls aged 18-60 years who included in the study. Of the cases at the beginning and at the end of the treatment; 5-10 cc peripheral blood samples were taken into one Ethylenediaminetetraacetic acid tube. Then Numeric Rating Scale (NRS) was used for pain, 28-joint Disease Activity Score (DAS28) was used to calculate disease activity, Health Assessment Questionnaire (HAQ) was used to assess general health and Short Form-36 (SF-36) was used to evaluate quality of life. In the samples taken, gene expressions of miRNA-146a, miRNA-155, miRNA-16, miRNA-145 were determined by real-time polymerase chain reaction method.
  Interventions: Behavioral: exercise; Biological: gene expressions of miRNA

INTERVENTIONS:
Behavioral: exercise — A program consisting of strengthening and stretching exercises 2 days a week was applied to the study group for 8 weeks. One day a week, 30 minutes of mild moderate walking was requested.
Biological: gene expressions of miRNA — In the samples taken, gene expressions of miRNA-146a, miRNA-155, miRNA-16, miRNA-145 were determined by real-time polymerase chain reaction method.

SUMMARY:
The goal of this prospective cohort study is to learn about whether exercise alters microRNA expression levels in 30 rheumatoid arthritis patients and 30 healthy controls.

The main questions it aims to answer are:

* Does exercise affect microRNA expression levels related to the pathophysiology of rheumatoid arthritis?
* Are microRNA levels correlated with disease activity? Participants was applied program consisting of strengthening and stretching exercises 2 days a week for 8 weeks. One day a week, 30 minutes of mild moderate walking was requested.

Researchers will compare rheumatoid arthritis patients and healthy controls to see if that the microRNA expression levels of patients with rheumatoid arthritis as a result of exercise training would not make a significant difference with healthy controls.

DETAILED DESCRIPTION:
Rheumatoid arthritis can be a systemic, inflammatory, autoimmune breathing that can cause heavy, joint destruction with vibrations in the synovial vessels of the joints. Although great strides have been made in understanding the disease, the pathogenesis of Rheumatoid arthritis.A has not yet been fully elucidated. Early treatment can prevent serious disability.

The goal of treatment for patients with rheumatoid arthritis is to achieve remission or at least a state of low disease activity.Combinations with disease-modifying antirheumatic drugs (DMARDs) and biologic agents are recommended for patients who fail to respond to treatment, based on patient prognosis and response to treatment.

In addition to drug therapy, exercise training is recommended in patients with Rheumatoid arthritis. Decreased joint health, including joint pain and inflammation, fatigue, increased incidence of cardiovascular disease in patients with rheumatoid arthritis; it causes functional limitation, disability, comorbidities and a decrease in quality of life.Therefore, it is recommended that aerobic and resistance exercise training should be encouraged as part of the routine treatment of all Rheumatoid arthritis patients.

microRNAs (miRNAs) are small, non-coding RNAs that mediate messenger RNA (mRNA) cleavage, translational repression. As regulators of gene expression, miRNAs participate in critical cellular processes and show varying levels of expression in many cell types in different diseases.It became clear that there were changes in miRNA expression in Rheumatoid arthritis patients.In many studies, it has been shown that miRNAs contribute to the disruption of joint destruction, inflammation and apoptosis in peripheral blood mononuclear cells, isolated T lymphocytes, synovial tissue and synovial fibroblasts. Thus, miRNAs are known to constitute the pathophysiological process specific to Rheumatoid arthritis.

miRNA-146a is one of the miRNAs that has been extensively studied in Rheumatoid arthritis. It was found that the expression of miRNA-146a in the synovial fluid and synovial tissue of Rheumatoid arthritis A patients was significantly higher than in healthy individuals, and miRNA-16 and miRNA-155 together with miRNA-146a may be related to disease pathology. In addition, high levels of miRNA-16 expression are known to correlate with active disease and low expression levels with remission. It has been reported that the expression level of miRNA-145 is increased in peripheral blood mononuclear cells and synovium of Rheumatoid arthritis patients, which supports osteoclastogenesis.

In this study, it was aimed to determine whether miRNAs, which play a role in determining the effectiveness of the treatment and the severity of the disease, change with exercise training, to know the effect of exercise training on the person, to accept it as an auxiliary practice in controlling the disease and to prove it with scientific facts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with not having any deformity in the last six months, not having a diagnosed cardiovascular disease

Exclusion Criteria:

* Exclusion criteria were not giving written consent, severe hypertension that would prevent physical activity, orthopedic problems that would prevent participation in the study, uncontrolled chronic systemic disease, central and peripheral nervous system diseases, recent neurological, orthopedic or other

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Pre-Treatment DAS28 for Treatment Group | Baseline
  28-joint Disease Activity Score (DAS28), which is widely used in clinics, is used to find disease findings in patients with rheumatoid arthritis. Calculation is made with the C-Reactive Protein value. DAS28> 5.1 is considered high disease activity, 3.2<DAS28≤5.1 is considered moderate disease activity, DAS28≤3.2 is low disease activity, and DAS28<2.6 is considered disease remission.
Post-Treatment DAS28 for Treatment Group | Through study completion, an average of 2 months
  28-joint Disease Activity Score (DAS28), which is widely used in clinics, is used to find disease findings in patients with rheumatoid arthritis. Calculation is made with the C-Reactive Protein value. DAS28> 5.1 is considered high disease activity, 3.2<DAS28≤5.1 is considered moderate disease activity, DAS28≤3.2 is low disease activity, and DAS28<2.6 is considered disease remission.
Pre-Treatment Gene Expressions of microRNA for Treatment Group | Baseline
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.
Post-Treatment Gene Expressions of microRNA for Treatment Group | Through study completion, an average of 2 months
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.
Gene Expressions of microRNA for Healthy Control Group | Baseline
  By examining the expression level of RNA, U6 small nuclear 1 (human) as a control gene, it is decided whether the expression levels of microRNAs are expressed up or down.

SECONDARY OUTCOMES:
NRS | at the beginning of the intervention and through study completion, an average of 2 month
  Then Numeric Rating Scale (NRS) was used for pain. In this scale, pain intensity is measured with an 11-point scale. Here 0: No pain and 10: the most severe pain level.
HAQ | at the beginning of the intervention and through study completion, an average of 2 month
  Health Assessment Questionnaire was used to assess general health. It consists of 20 questions in total, including 8 subsections. Subjects score between 0-3 according to their level of difficulty in activities. The total score is obtained by calculating the arithmetic mean of the sums of the highest scores in the subsections. Higher scores indicate higher functional disability and pain.
SF-36 | at the beginning of the intervention and through study completion, an average of 2 month
  Short Form-36 (SF-36) was used to evaluate quality of life. This Questionnaire consists of eight subsections. Scoring is made between 0-100 for each of the subsections. Higher scores indicate better function and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Betül ÖZCAN, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Fulya Senem KARAAHMETOĞLU, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Bekir ERDOĞAN, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Sibel KURAŞ, M. Sc., Study Chair — Saglik Bilimleri Universitesi; Mehmet Zahid ÇIRACI, MD, Principal Investigator — Sakarya Training and Research Hospital; Halime Hanım PENÇE, Assoc. Pr, Study Chair — Saglik Bilimleri Universitesi; Meltem VURAL, Prof. Dr., Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospital; Alev KURAL, Assoc. Pr., Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospital; Işıl ÜSTÜN, MD, Study Chair — Istanbul Bakırköy Dr.Sadi Konuk Training and Research Hospital
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Turkey (Türkiye)